CLINICAL TRIAL: NCT01725230
Title: An Open-label, Non-randomized, 2-Period, Fixed Sequence, Single-center Study to Assess the Pharmacokinetics of Rosuvastatin and Simvastatin in Healthy Subjects When Administered Alone and in Combination With Fostamatinib 100 mg Twice Daily
Brief Title: Assess the Pharmacokinetics of Rosuvastatin and Simvastatin When Administered Alone or in Combination With Fostamatinib
Acronym: Statin DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00039
Record Dates: First submitted 2012-11-07; First posted 2012-11-12 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Fostamatinib,; simvastatin,; rosuvastatin,; Phase I,; Healthy Subjects,; Pharmacokinetics
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib; Rosuvastatin Calcium; Simvastatin

ARMS (2):
- Rosuvastatin (Experimental): Single, oral dose of rosuvastatin 20mg in first period and in second period (after wash out) fostamatinib 100 mg twice daily, then single oral dose of rosuvastatin 20 mg plus continued oral dosing of fostamatinib 100 mg twice daily, then continue fostamatinib 100 mg twice daily
  Interventions: Drug: Fostamatinib; Drug: Rosuvastatin
- Simvastatin (Experimental): Single, oral dose of simvastatin 40 mg in first period and in second period (after wash out) fostamatinib 100 mg twice daily, then single oral dose of simvastatin 40 mg plus continued oral dosing of fostamatinib 100 mg twice daily, then continue fostamatinib 100 mg twice daily
  Interventions: Drug: Fostamatinib; Drug: Simvastatin

INTERVENTIONS:
Drug: Fostamatinib — 100-mg tablet
Drug: Rosuvastatin — 20-mg tablet
  Arms: Rosuvastatin
Drug: Simvastatin — 40-mg tablet
  Arms: Simvastatin

SUMMARY:
A study to Assess the Pharmacokinetics of Rosuvastatin and Simvastatin when administered alone or in combination with Fostamatinib.

DETAILED DESCRIPTION:
An Open-label, Non-randomized, 2-Period, Fixed Sequence, Single-center Study to Assess the Pharmacokinetics of Rosuvastatin and Simvastatin in Healthy Subjects when Administered Alone and in Combination with Fostamatinib 100 mg Twice Daily.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent, prior to any study-specific procedures
* Volunteers will be males or females aged 18 to 55 years and with a weight of at least 50 kg and body mass index (BMI) between 18 and 30 kg/m2, inclusive.
* Male volunteers should be willing to use barrier contraception, ie, condoms, from the day of first dosing until 2 weeks after the last dosing with IP.
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating, and must be of non childbearing potential, confirmed at screening .

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IP as judged by the Investigator.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the Investigator.
* Any clinically significant abnormal findings in vital signs as judged by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Rosuvastatin measured by AUC and Cmax. | Day 1 and Day 6 at predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours postdose.
Pharmacokinetics of Simvastatin measured by AUC and Cmax | Day 1 and Day 6 at predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours postdose.

SECONDARY OUTCOMES:
Pharmacokinetics of R406 measured by AUC(0-t), Cmax, Tmax (alone and in combination with rosuvastatin or simvastatin) | Day 1 to day 4 at predose, Day 5 and Day 6 at predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours postdose.
Pharmacokinetics of rosuvastatin measured by AUC(0-t), t1/2, Tmax, Cl/F and Vz/F (alone and in combination with fostamatinib) | Day 1 and Day 6 at predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours postdose.
Pharmacokinetics of Simvastatin measured by AUC(0-t)m t1/2, and Tmax (alone and in combination with fostamatinib) | Day 1 and Day 6 at predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours postdose.
Pharmacokinetics of simvastatin measured by AUC, Cmax, AUC(0-t), t1/2, Tmax, C1/F and Vz/F (alone and in combination with fostamatinib) | Day 1 and Day 6 at predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours postdose.
Frequency of adverse events | Measured throughout the study and 3-5 days after discharge from Period 2, approximately 72 days
Severity of adverse events | Measured throughout the study and 3-5 days after discharge from Period 2, approximately 72 days

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles Phase I unit 6700 w 115th st Overland Park, Ks 66211; Christopher D O'Brien, MD PHD, Study Director — AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States